CLINICAL TRIAL: NCT05771285
Title: The Effect of Cold Application on the Occurrence of Bruising, Hematoma and Pain in the Subcutaneous Low Molecular Weight Heparin Injection: a Randomized Controlled Trial
Brief Title: Cold Application on the Subcutaneous Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, cevahir ilkim buldak, Lecturer, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Cold App
Record Dates: First submitted 2022-12-22; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Injection Site Bruising; Bruising; Pain
Keywords: bruising; cold application; haematoma; low molecular weight heparin; nursing; pain; subcutaneous injection
MeSH Terms: conditions — Contusions; Pain; Hematoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group with two-minute pre-injection application of cold (Active Comparator): Before applying the subcutaneous injection, cold application pack was applied on the injection site for two minutes. Then, the low molecular weight heparin injection was applied to this cold-applied area in accordance with the subcutaneous heparin injection protocol. VAS assessment was made after the injection and bruise and haematoma assessments were conducted after 48 and 72 hours.
  Interventions: Other: Cold application
- Group with five-minute pre-injection application of cold (Active Comparator): Before applying the subcutaneous injection, cold application pack was applied on the injection site for five minutes. Then, the low molecular weight heparin injection was applied to this cold-applied area in accordance with the subcutaneous heparin injection protocol. VAS assessment was made after the injection and bruise and haematoma assessments were conducted after 48 and 72 hours.
  Interventions: Other: Cold application
- Control group (No Intervention): Without applying any tools or processes, the low molecular weight heparin injection was applied in accordance with the subcutaneous heparin injection protocol. VAS assessment was made after the injection and bruise and haematoma assessments were conducted after 48 and 72 hours.

INTERVENTIONS:
Other: Cold application — To evaluate the effect of cold application applied before subcutaneous low molecular weight heparin injection on post-injection pain, ecchymosis and hematoma formation.
  Arms: Group with five-minute pre-injection application of cold; Group with two-minute pre-injection application of cold

SUMMARY:
The goal of this clinical trial is to compare the effect of cold application at different periods of time on the occurrence of bruising, haematoma and pain in the subcutaneous low molecular weight heparin (LMWH) injected patients.

DETAILED DESCRIPTION:
The study was a single-blind randomised control trial. Patients were allocated randomly to three groups: (i) Cold was applied for two minutes before the injection in the first group (n=26); (ii) Cold was applied for 5 min before the injection in the second group (n=26); and (iii) control group (n=26). All participating patients were injected 40 mg enoxaparin sodium in 0.4 ml in the pre-filled syringes using standard LMWH injection protocol. Post-injection VAS (Visual Analogue Scale) assessment and assessment of the presence and size of bruise and haematoma were conducted at 48th and 72nd hours after the injections for all groups.

ELIGIBILITY:
Inclusion Criteria:

* to receive LMWH (pre-filled syringe containing 40 mg enoxaparin sodium in 0.4 ml) treatment at least once a day
* not to have any visual or auditory disorders
* not to have any foreknown coagulation disorders
* to have platelet, PTT and international normalized ratio (INR) values within the normal limits for beginning enoxaparin sodium injections
* not to have any hematologic disorders or any bruising or injuries at the abdominal wall
* to receive no injections at the abdominal site, other than the enoxaparin sodium during the research protocol
* to will to participate in this study

Exclusion Criteria:

* to be pregnant
* have bleeding in the injection site
* have pain at any site of their body prior to the injection
* have any incision, drain, scar tissue, lipodystrophy or infection symptoms at the abdominal site which hinder the application of injection
* not to will to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Compare of the bruise occurrence change at 48th and 72nd hours after the heparin injection. | after 48th and 72nd hours from injection
  It was evaluated whether bruise occurred 2 times at 48th and 72nd hours after heparin injection.
Compare of the bruise sizes change of the patients at 48th and 72nd hours. | after 48th and 72nd hours from injection
  If bruise developed after heparin injection, its size was measured 2 times at 48th and 72nd hours and recorded.
Compare of the Visual Analogue Scale pain scores of the patients | after 1 minute from injection administration
  The level of pain felt after the heparin injection administration was measured with the visual analogue scale. Visual Analogue Scale (VAS) was used to measure the extent of pain during the injection. VAS is widely used to measure the clinical symptoms such as pain, panic, depression, and fatigue. VAS consists of 100 mm on a horizontal line. On the scale "0" means no pain and "100" shows severe pain. The patients were asked to mark the extent of pain they had immediately after the subcutaneous injection on the scale with 'X'. The distance from "no pain" to the place that the patient has marked quantitatively represents the pain of the patient.

SECONDARY OUTCOMES:
Occurrence of haematoma at 48th and 72nd hours after the heparin injection. | after 48th and 72nd hours from injection
  Changes in hematoma formation were evaluated at 48 and 72 hours after heparin injection.

CONTACTS AND LOCATIONS:
Overall Officials: Cevahir İlkim BULDAK, Principal Investigator — ilkimbuldak@yiu.edu.tr